CLINICAL TRIAL: NCT06149611
Title: Clinical Study on Material Balance of [14C]TQB3616 in Healthy Chinese Subjects
Brief Title: Mass Balance Study of TQB3616
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TQB3616-I-04
Record Dates: First submitted 2023-11-21; First posted 2023-11-29 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- [14C] TQB3616 (Experimental): 100 µCi [14C] TQB3616, 180mg, once in total.
  Interventions: Drug: [14C] TQB3616

INTERVENTIONS:
Drug: [14C] TQB3616 — TQB3616 is a new type of cyclin-dependent kinase (CDK) 4/6 inhibitor.

SUMMARY:
This is a clinical study exploring the mass balance of [14C] TQB3616 in healthy Chinese subjects aims to quantitatively analyze the total radioactivity in the feces of male healthy subjects after oral administration of [14C] TQB3616, obtain data on human radiation excretion rate and main excretion pathways, investigate the distribution in whole blood and plasma, plasma distribution, and pharmacokinetics of total radioactivity in plasma, identify main metabolites, and determine the main biological transformation pathways, obtain the pharmacokinetic parameters of TQB3616 and its metabolites in plasma. The primary endpoint is mass balance, radiopharmacokinetics, plasma pharmacokinetics, and metabolites.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult male;
* Age: 18-45 years old (inclusive);
* The body mass index (BMI) is between 19-26 kg/m2 (inclusive), and the subject's body weight shall be not less than 50 kg (inclusive);
* Voluntarily sign the informed consent form;
* The subjects are able to communicate well with the investigators and complete the study according to the protocol.

Exclusion Criteria:

* Abnormal and clinically significant results in comprehensive physical examination, vital signs, digital examination of the anus, laboratory examination (blood routine, blood biochemistry, urine routine, coagulation function, fecal routine+occult blood, thyroid function, etc.), 12-lead electrocardiogram, chest X-ray (Posterior-anterior), abdominal ultrasound (liver, gallbladder, pancreas, spleen, kidney), ect.;
* Abnormal and clinically significant results in ophthalmic examinations (slit lamp, intraocular pressure, and fundus photography);
* Any one of hepatitis B surface antigen, hepatitis B e antigen, hepatitis C antibody, HIV antibody and syphilis antibody is positive;
* Within 30 days before the screening period, those who have used any drugs that inhibit or induce liver drug metabolism (such as CYP3A4 inducers like carbamazepine, dexamethasone, rifampicin, phenytoin, phenobarbital, rifabutin, rifapentine, hypericum perforatum, etc.; CYP3A4 inhibitors like itraconazole, ketoconazole, clarithromycin, voriconazole, telithromycin, saquinavir, lopinavir, ritonavir, etc.);
* Within 14 days prior to the screening period, have taken any prescription drugs, over-the-counter drugs, Chinese herbal medicines, or health products;
* Those who have participated in any drug clinical trial and received any investigational drug within 3 months prior to the screening period;
* Have a history of any clinically serious illness or condition that the investigator believes may affect the test results, including but not limited to a history of circulatory, endocrine, nervous, digestive, urinary, or blood, immune, mental, and metabolic diseases;
* Having undergone major surgery or incomplete healing of the surgical incision within 6 months prior to the screening period; Major surgeries include, but are not limited to, any surgeries with significant bleeding risks, prolonged general anesthesia, or open biopsies or obvious traumatic injuries.
* Individuals with allergic constitution, including those with a history of drug allergy, known to be allergic to TQB3616 or similar drugs or its excipients, be allergic to any food ingredient or has special dietary requirements, and cannot follow a unified diet;
* Hemorrhoids or perianal diseases with regular/ongoing bloody stools; The presence of gastrointestinal dysfunction such as irritable bowel syndrome and inflammatory bowel disease that may affect drug absorption, distribution, metabolism, and excretion, as determined by investigators;
* Habitual constipation or diarrhea;
* Excessive drinking or frequent drinking within 6 months prior to the screening period, i.e. drinking more than 14 units of alcohol per week (1 unit=360 mL of beer or 45 mL of 40% alcohol or 150 mL of wine); Or during the screening period, the alcohol breath test result is ≥ 20 mg/dL;
* Those who smoke more than 5 cigarettes per day or habitually use nicotine containing products within 3 months prior to the screening period, and are unable to quit during the trial period;
* Abuse of drugs or use of soft drugs (such as marijuana) within 3 months prior to the screening period, or use of hard drugs (such as cocaine, amphetamines, phencyclidine, etc.) within 1 year prior to the screening period; Positive urine drug abuse test during screening period;
* Habitually drinking grapefruit juice or excessive amounts of tea, coffee, and/or caffeinated beverages, and unable to quit during the study period;
* Engaged in working that require long-term exposure to radioactive conditions; Or those who have significant radiation exposure (≥ 2 chest/abdominal CT scans, or ≥ 3 other types of X-ray examinations) or participated in radiopharmaceutical labeling tests within 1 year before the study;
* Those who have received vaccines within 1 month before screening or have vaccination plans during the study;
* Individuals with a history of needle or blood fainting and have difficulty or cannot tolerate venous puncture for blood collection;
* Those who have fertility plans during the study period and within 1 year after the completion of the study; or those who do not agree to adopt strict contraceptive measures during the experiment and within 1 year after the completion of the study;
* Individuals who have experienced blood loss or donated up to 400 mL of blood within 3 months prior to the screening period, or have received blood transfusions, or plan to donate blood within 1 month after the end of this study;
* Subjects that are not suitable for participating in this study due to other factors as judged by the investigators.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Estimated)
Dates: Start 2024-01 (Estimated); Primary Completion 2024-06 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Peak concentration (Cmax) | Pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 24, 48, 72, 96, 120, 144, 168, 216, 264, 336 hours after dose.
  Maximum plasma drug concentration
Area under drug time curve | Pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 24, 48, 72, 96, 120, 144, 168, 216, 264, 336 hours after dose.
  Area under the blood concentration time curve
Time to peak concentration (Tmax) | Pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 24, 48, 72, 96, 120, 144, 168, 216, 264, 336 hours after dose.
  Time to reach maximum (peak) plasma concentration following drug administration
Elimination half-life (t1/2) | Pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 24, 48, 72, 96, 120, 144, 168, 216, 264, 336 hours after dose.
  The time it takes for the blood concentration of a drug to decrease from its highest value to half in the body.
Mean resident time (MRT) | Pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 24, 48, 72, 96, 120, 144, 168, 216, 264, 336 hours after dose.
  The average time that drug molecules remain in the body.

SECONDARY OUTCOMES:
Adverse event rate | Baseline up to 21 days after administration
  The incidence of adverse events after administration.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu, China